## Efficacy of Dry Needling in Plantar Fasciitis

NCT number: 02467465

Madrid, 23th april 2014.

## STATISTICAL METHOD:

Initially, a descriptive statistical analysis will be carried out: the qualitative variables will be summarized by the frequency and percentage distribution, and the quantitative variables by their mean and standard deviation. Likewise, the information will be summarized graphically by means of box plots and sector graphs.

In addition, the Shapiro Wilk test will be carried out to test the normality of the sample. From this result, the inferential analysis will be made using parametric or non-parametric techniques. In particular, to assess the differences in the pre- and post-intervention responses, the average range test will be used with the Wilcoxon test (in cases of a normal distribution for the response variable) or the Student's t-test for related samples. For the study of the response variables between groups, the Mann-Whitney U test and the Student t test for independent samples will be used.

For all these tests, significant differences are assumed in values of p <0.05 and a confidence interval of 95%. The statistical analysis will be carried out through the Statistical Software SPSS v19.0.